CLINICAL TRIAL: NCT00405067
Title: A Randomized, Double-Blind, Active Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of the Combination BMS-201038 (AEGR-733) and Ezetimibe vs. Monotherapy in Subjects With Moderate Hypercholesterolemia
Brief Title: The Safety & Efficacy of Combination BMS-201038 (AEGR-733) & Ezetimibe vs. Monotherapy in Moderate Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEGR-733-001
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — BMS201038; Ezetimibe

INTERVENTIONS:
Drug: BMS-201038 (AEGR-733)
Drug: Ezetimibe

SUMMARY:
The main objectives of this study are to evaluate the efficacy and safety of combination therapy BMS-201038 (AEGR-733) plus ezetimibe vs. each agent given alone on LDL cholesterol and other lipoproteins over 12 weeks of therapy.

DETAILED DESCRIPTION:
Subjects will participate in this study for approximately 14-17 weeks. This study has 2 periods: 1) a 1-2-week screening period with 2 visits where baseline cholesterol and other characteristics will be evaluated to determine study eligibility. This period also includes a 4-week washout for patients on prior lipid-lowering therapies; and 2) a 12-week treatment period with interim visits at weeks 4 and 8.

85 subjects were randomized into one of 3 treatment arms with equal probability. In treatment arm 1, subjects will receive BMS-201038 (AEGR-733) 5 mg plus ezetimibe placebo. In treatment arm 2, subjects will receive BMS-201038 (AEGR-733) placebo plus 10 mg of ezetimibe. In treatment arm 3, subjects will receive BMS-201038 (AEGR-733) 5 mg plus ezetimibe 10 mg. After 4 weeks of treatment, subjects in arms 1 and 3 will be force-titrated to BMS-201038 (AEGR-733) 7.5 mg. After another 4 weeks of treatment, subjects in arms 1 and 3 will then be force-titrated to BMS-201038 (AEGR-733) 10 mg for 4 more additional weeks of treatment. Subjects in arm 2 will continue to receive BMS-201038 (AEGR-733) matching placebo for the entire 12 weeks of treatment. Subjects randomized to ezetimibe 10 mg in arms 2 and 3 and ezetimibe placebo in arm 1 will remain on these doses for the entire 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 70 years .
2. For subjects with 0 to 1 risk factor (cigarette smoking, hypertension (BP > 140/90 or on antihypertensive medication), low HDL (<40mg/dl), family history of premature CHD (CHD in male first degree relative <55 years; CHD in female first degree relative <65 years), age (men> 45 years; women > 55 years): Baseline mean LDL-C must be >160 and <250 mg/dl as determined by the arithmetic mean of measures taken at visit 1 and 2. Fasting mean TGs should be <400 mg/dl.
3. For subjects with 2 or more risk factors (cigarette smoking, hypertension (BP > 140/90 or on antihypertensive medication), low HDL (<40mg/dl), family history of premature CHD (CHD in male first degree relative <55 years; CHD in female first degree relative <65 years), age (men> 45 years; women > 55 years) or prior stable CHD: Baseline mean LDL-C must be >130 and <250 mg/dl as determined by the arithmetic mean of measures taken at visit 1 and 2. Fasting mean TGs should be <400 mg/dl.
4. Able to understand and willing to comply with all study requirements, particularly the study drug regimen.
5. Able to understand and willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Women who are pregnant or lactating or who are planning to become pregnant or women of child bearing potential who have not successfully been using acceptable contraceptive methods over the previous 3 months (e.g. intrauterine device and barrier method plus spermicide).
2. Uncontrolled hypertension defined as: systolic blood pressure > 180 mmHg, diastolic blood pressure > 95 mmHg
3. History of chronic renal insufficiency (serum creatinine >2.5 mg/dL)
4. History of liver disease or transaminases above 1.5 X ULN at screening
5. Any major surgical procedure occurring less than 3 months prior to the screening visit
6. Cardiac insufficiency defined by the NYHA classification as functional Class II-Class IV
7. History of a malignancy (other than basal cell or squamous cell carcinoma of the skin that has been removed) within the previous 5 years
8. Participation in an investigational drug study within 6 weeks prior to the screening visit.
9. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
10. Regular alcohol use > 1 drink per day
11. Regular consumers of grapefruit juice, or currently taking medications known to be metabolized by CYP 3A4 (cyclosporine, itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, and nefazodone)
12. Other lipid-lowering medications (washouts will be permitted)
13. Acute CVD (CVD event within the previous 6 months)
14. Diabetes Mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davidson, MD, Principal Investigator — Radiant Research; Jackson Downey, MD, Principal Investigator — Jacksonville Center For Clinical Research; Paul Grena, MD, Principal Investigator — Cardiology Consultants of Philadelphia; Barry Lubin, MD, Principal Investigator — Hampton Roads Center for Clinical Research; James McKenney, Pharm D, Principal Investigator — National Clinical Research; Eli Roth, MD, Principal Investigator — Sterling Research Group, LTD
Locations (1):
- Pharmanet, Inc, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed from 30 Jun 2006 to 27 Dec 2006. A total of 6 medical clinics participated in the study.
Pre-assignment Details: Patients who were previously on a lipid lowering therapy underwent a 4-week washout period.
Groups:
- Combination Therapy: Oral ezetimibe 10 mg and lomitapide escalated with an initial oral dose of 5 mg for 4 weeks and then escalated through 2 additional dose levels (7.5 mg and 10 mg) every 4 weeks over an 8-week period.
- Lomitapide Monotherapy: Oral ezetimibe placebo and lomitapide escalated with an initial oral dose of 5 mg for 4 weeks and then escalated through 2 additional dose levels (7.5 mg and 10 mg) every 4 weeks over an 8-week period.
- Ezetimibe Monotherapy: Oral ezetimibe 10 mg and lomitapide placebo for 12 weeks.
Period: Overall Study
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Started | 28 | 28 | 29
Completed | 24 | 19 | 24
Not Completed | 4 | 9 | 5
Not completed — Adverse Event | 4 | 9 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy | Total
Number analyzed (Participants) | 28 | 28 | 29 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (5.7) | 57.5 (7.2) | 54.7 (9.0) | 55.7 (7.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 18 | 45
  Male | 14 | 15 | 11 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 6 | 7 | 22
  White | 18 | 22 | 22 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 29 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in LDL-C at 12 Weeks Therapy Compared to Baseline Between Treatments
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 19 | 24
Percent Change | -46.2 (23.8) | -29.9 (15.3) | -19.6 (9.9)

2. Secondary Outcome: Percent of Change at 12 Weeks Therapy Compared to Baseline Between Treatments for the Following Parameters: Total Cholesterol (TC)
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 19 | 24
Percent Change | -34.4 (18.8) | -22.8 (12.3) | -12.0 (8.7)

3. Secondary Outcome: Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) at 12 Weeks as Compared to Baseline.
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 19 | 24
Percent Change | -41.3 (22.7) | -26.9 (14.6) | -17.0 (10.5)

4. Secondary Outcome: Percent Change in Tryglycerides (TGs) at 12 Weeks Compared to Baseline
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 19 | 24
Percent Change | -7.0 (36.0) | -5.8 (33.6) | 2.7 (35.1)

5. Secondary Outcome: Percent Change in HDL-C at 12 Weeks Compared to Baseline
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 19 | 24
Percent Change | -9.2 (14.4) | -6.2 (10.8) | 5.9 (9.6)

6. Secondary Outcome: Percent Change in Lipoprotein(a)[Lp(a)]at 12 Weeks as Compared to Baseline
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 20 | 18 | 21
Percent Change | -12.0 (23.7) | -11.4 (29.1) | 7.5 (24.1)

7. Secondary Outcome: Percent Change in Apolipoprotein A1 (Apo A1) at 12 Weeks as Compared to Baseline
Time Frame: baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 18 | 23
Percent Change | -10.7 (15.8) | -8.0 (12.3) | 2.3 (9.5)

8. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B) at 12 Weeks as Compared to Baseline
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 18 | 23
Percent Change | -36.6 (21.7) | -23.7 (14.2) | -14.5 (10.6)

9. Secondary Outcome: Percent Change in High-sensitivity C-reactive Protein (Hs-CRP) at 12 Weeks as Compared to Baseline
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 19 | 24
Percent Change | 40.4 (80.7) | 81.3 (337.6) | 233.3 (874.9)

10. Secondary Outcome: Percent Change in Body Weight at 12 Weeks as Compared to Baseline
Time Frame: Baseline and 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Number analyzed (Participants) | 24 | 19 | 24
Percent Change | -1.4 (2.9) | -1.0 (2.2) | -0.1 (2.3)

ADVERSE EVENTS:
Arm/Group | Combination Therapy | Lomitapide Monotherapy | Ezetimibe Monotherapy
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/28 | 0/29
Other Adverse Events (participants affected / at risk) | 24/28 | 24/28 | 15/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=28) | Lomitapide Monotherapy (N=28) | Ezetimibe Monotherapy (N=29)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=28) | Lomitapide Monotherapy (N=28) | Ezetimibe Monotherapy (N=29)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 11 (11) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (5) | 8 (8) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 7 (7) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Liver function test abnormal (Investigations) | 3 (3) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after sponsor has 60 days to review the proposed publication. PI is committed to publish the results of the study in a cooperative publication with other investigators prior to individual publication. PI needs sponsor's prior consent to publish confidential information, not to be unreasonably withheld. The PI shall, upon sponsor's request, delete from the publication any confidential information which would prejudice the securing of adequate intellectual property protection.